CLINICAL TRIAL: NCT05006196
Title: Contrast-Free Magnetic Resonance Imaging for Breast Disease
Acronym: IMOGEN
Status: Active, not recruiting | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: 20/WS/0110
Record Dates: First submitted 2021-07-14; First posted 2021-08-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Breast Diseases
Keywords: Breast imaging; Magnetic resonance imaging; Screening
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Genotype; Body Height; Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The tests consist of complete blood count (CBC), biochemical profile and stored serum/plasma. Genetic testing for genetic variants associated with this disease may also be carried out if the participant gives informed consent for genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Outpatient MRI — Participation in the study includes up to a maximum of 2 study visits. The visits will include clinical measurements (height, weight, blood pressure), blood tests, MRI scan and patient symptoms and experience questionnaires.
  There will be no medical interventions as part of the study. All participants will receive standard-of-care by their healthcare provider/s. With the participant's consent, the participant's primary care physician will be made aware of their participation in the study. Furthermore, participants will be informed of any structural abnormalities found in the MRI scan (e.g. abnormal vessels, haemangioma, tumour, cyst, among others) and abnormal blood test results as these may have clinical implications. These will be managed by the routine clinical care team as part of standard care.
  Other Names: Outpatient blood tests for laboratory studies and genotyping; Outpatient measurements (height, weight, blood pressure); Patient questionnaires

SUMMARY:
Prospective, observational cohort study looking at patients either at risk of breast cancer or have clinically suspected breast to assess the diagnostic performance of quantitative, non-contrast MRI.

DETAILED DESCRIPTION:
It is widely recognised that mammography is highly sensitive for detecting breast lesions and a valuable tool for early detection of breast cancer, especially in post-menopausal women with non-dense breast tissue. On post-menopausal non-dense breast tissue, mammography is 90% effective at identifying breast tumours. However, for dense breast tissue, the sensitivity falls to 67%. This means that for women with dense breast tissue, which includes almost all pre-menopausal women and many post- menopausal women, mammography misses one third of tumours.

MRI is the imaging method of choice for detecting breast cancer in women with dense breast tissue however the standard MRI for breast cancer investigation typically uses gadolinium contrast agent. This method is called dynamic contrast enhanced (DCE) MRI and identifies localised regions of (neo)vascularity, which indicates a cancerous lesion. Although DCE can provide valuable information about the tissue, it is often not performed well, is poorly tolerated by patients, and adds additional time to the scan protocol.

Perspectum conducted a recent study demonstrating that liver cancer lesions can be identified using quantitative T1 maps calculated form multiparametric MRI data. Applying this MRI method to breast imaging, would potentially provide a method of identifying breast cancer lesions without using a contrast agent, reducing the scan time and eliminating the need for an intravenous contrast.

The aim of this study is to apply quantitative multiparametric MRI techniques to the area of breast imaging with the aim of developing a contrast-free MR scan which can diagnose the spectrum of breast disease referred to a secondary care breast clinic, including in women with dense breasts.

ELIGIBILITY:
Inclusion Criteria:

* Female 30 years of age and over
* Participant has been referred to a secondary care breast screening clinic.
* Participant is willing and able to give informed consent for participation in the investigation.

Exclusion Criteria

* The participant may not enter the study with any known contraindication to magnetic resonance imaging (including but not limited to a pacemaker or other metallic unfixed implanted device, metallic fragments, extensive tattoos, severe claustrophobia).
* Any other cause, including a significant underlying disease or disorder which, in the opinion of the investigator, may put the participant at risk by participating in the study or limit the participant's ability to participate.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women at risk of breast cancer or who have suspected breast disease aged 30 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 1030 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Determine the diagnostic performance of a non-contrast MRI in breast disease | 36 months
  Mapping multi-parametric algorithms and assessing diagnostic performance compared to standard of care using area under the receiver operative curve (AUROC)

SECONDARY OUTCOMES:
Qualitatively assess the participant experience of identifying breast disease using non-contrast MRI | 36 months
  Provide participants with a non validated questionnaire and summarise feedback on MR techniques compared to standard of care

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, MSc, DPhil, Principal Investigator — Honorary Consultant Physician, Oxford University NHS Foundation Trust
Locations (1):
- Gemini One, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At the end of the study, the pooled and anonymous results of the questionnaires will be available to all participants upon their request. No individual participant will be identified.

REFERENCES:
- [Background] von Euler-Chelpin M, Lillholm M, Vejborg I, Nielsen M, Lynge E. Sensitivity of screening mammography by density and texture: a cohort study from a population-based screening program in Denmark. Breast Cancer Res. 2019 Oct 17;21(1):111. doi: 10.1186/s13058-019-1203-3. PMID 31623646
- [Background] Bakker MF, de Lange SV, Pijnappel RM, Mann RM, Peeters PHM, Monninkhof EM, Emaus MJ, Loo CE, Bisschops RHC, Lobbes MBI, de Jong MDF, Duvivier KM, Veltman J, Karssemeijer N, de Koning HJ, van Diest PJ, Mali WPTM, van den Bosch MAAJ, Veldhuis WB, van Gils CH; DENSE Trial Study Group. Supplemental MRI Screening for Women with Extremely Dense Breast Tissue. N Engl J Med. 2019 Nov 28;381(22):2091-2102. doi: 10.1056/NEJMoa1903986. PMID 31774954
- [Background] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764